CLINICAL TRIAL: NCT00050011
Title: An Open-Label, Randomized, Multicenter Study to Evaluate the Use of Zoledronic Acid in the Prevention of Cancer Treatment-Related Bone Loss in Postmenopausal Women With Estrogen Receptor Positive and/or Progesterone Receptor Positive Breast Cancer Receiving Letrozole as Adjuvant Therapy
Brief Title: Zoledronic Acid - Letrozole Adjuvant Synergy Trial (ZFAST) - Cancer Treatment Related Bone Loss in Postmenopausal Women With Estrogen Receptor Positive and/or Progesterone Receptor Positive Breast Cancer Receiving Adjuvant Hormonal Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CZOL446EUS32
Record Dates: First submitted 2002-11-18; First posted 2002-11-20 (Estimated); Results first posted 2014-01-28 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-02

CONDITIONS: Breast Neoplasms; Osteoporosis
Keywords: cancer-treatment related bone loss; postmenopausal women; breast cancer; hormone receptor positive breast cancer; adjuvant therapy; hormonal therapy; bone loss; bisphosphonates; ZFAST; Letrozole; Zoledronic Acid; US32
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis; Bone Diseases, Metabolic | interventions — Zoledronic Acid; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zoledronic Acid upfront (Experimental): Participants in the upfront arm received zoledronate 4 mg i.v. on Day 1 and every 6 months until disease progression (recurrence) or the end of study. Participants also received Letrozole 2.5 daily plus calcium (1000-1200 mg) and vitamin D (400-800 IU) daily.
  Interventions: Drug: Zoledronic Acid; Drug: Letrozole
- Zoledronate delayed-start (Experimental): In lieu of a placebo arm, which was considered unethical for this trial, a delayed start arm was used. Participants who met certain clinical criteria indicating risk of lumbar spine or total hip fracture, or experienced clinical fracture unrelated to trauma or any asymptomatic fracture discovered at the Month 36 scheduled visit, were started on zoledronate 4 mg i.v. and for every 6 months until disease progression (recurrence) or end of study. Participants also received Letrozole 2.5 daily plus calcium (1000-1200 mg) and vitamin D (400-800 IU) daily.
  Interventions: Drug: Zoledronic Acid; Drug: Letrozole

INTERVENTIONS:
Drug: Zoledronic Acid — Participants received Zoledronate 4 mg IV 15-minute infusion every 6 months.
  Other Names: ZOL446; Zoledronate
Drug: Letrozole — Participants received Letrozole 2.5 mg daily.
  Other Names: Femara

SUMMARY:
This protocol is designed to compare the effect on bone of Zoledronic Acid 4 mg every 6 months when given upfront versus delayed start (based on a post-baseline BMD T- Score below -2.0 SD at either the lumbar spine or total hip, or any clinical fracture unrelated to trauma, or an asymptomatic fracture discovered at the month 36 scheduled visit) in stage I-IIIb postmenopausal women with hormone receptor positive breast cancer who will receive Letrozole 2.5 mg daily as an adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Postmenopausal status defined by one of the following :

   * women equal to or greater than 55 years with cessation of menses
   * spontaneous cessation of menses within the past 1 year, but amenorrheic in women less than or equal to 55 years (e.g., spontaneous or secondary to hysterectomy), and with postmenopausal gonadotrophin levels (follicle stimulating hormone levels >40 IU/L) or postmenopausal estradiol levels (< 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved
   * bilateral oophorectomy (prior to the diagnosis of breast cancer).
3. Adequately diagnosed and treated breast cancer defined as:

   * Patients with breast cancer whose tumor can be removed by an appropriate surgical procedure such as mastectomy or breast conserving surgery and who receive appropriate additional local treatments such as radiotherapy according to best practice.
   * Patients must be at the end of their local treatment without evidence of local residual disease.
   * Patients must have no clinical or radiological evidence of distant metastasis.
4. Hormone receptor positive defined as:

   * ER and/or PR greater than or equal to1 0 fmol/mg cytosol protein; or greater than or equal to 10% of the tumor cells positive by
   * immunohistochemical evaluation.
5. Patients with a baseline lumbar spine and total hip BMD T-score at or above -2.0 SD are eligible.
6. Patients who will receive adjuvant chemotherapy are eligible for participation. Adjuvant chemotherapy must be completed prior to randomization.
7. The date of randomization must not be more than the following:

   * 12 weeks from completion of surgery;
   * 12 weeks after completion of adjuvant chemotherapy;
   * 12 weeks after completion of surgery and radiation therapy; however the patient may be randomized while receiving radiation therapy - this decision is at the Investigator's discretion.
   * 12 weeks after completion of chemotherapy and radiation therapy; however, the patient may be randomized while receiving radiation therapy - this decision is at the Investigator's discretion.
8. Patients who have undergone neoadjuvant chemotherapy are eligible.
9. No prior treatment with Femara.

Exclusion criteria:

1. Patients with any clinical or radiological evidence of distant spread of their disease at any point before randomization.
2. Patients with clinical or radiological evidence of existing fracture in the lumbar spine and/or total hip.
3. Patients with a history of fracture with low-intensity or no associated trauma.
4. Patients who have started adjuvant hormonal therapy or who have completed adjuvant hormonal therapy prior to randomization.
5. Patients who have received any endocrine therapy within the past 12 months (other than neoadjuvant tamoxifen or toremifene, insulin and/or oral anti-diabetic medications, and thyroid hormone replacement). Hormone replacement therapy must be discontinued prior to randomization.
6. Patients who have received prior treatment with intravenous bisphosphonates within the past 12 months.
7. Patients currently receiving oral bisphosphonates. Oral bisphosphonates must be discontinued within 3 weeks of baseline evaluations.
8. Patients who have received prior treatment with systemic corticosteroids within the past 12 months (short term corticosteroid therapy, e.g. to prevent/treat chemotherapy-induced nausea/vomiting, is acceptable).
9. Patients with prior exposure to anabolic steroids or growth hormone within the past 6 months.
10. Patients with prior use of Tibolone within the last 6 months.
11. Any prior use of PTH for more than 1 week.
12. Prior use of systemic sodium fluoride for > 3 months during the past 2 years.
13. Patients currently treated with any drugs known to affect the skeleton (e.g., calcitonin, mithramycin, or gallium nitrate) within 2 weeks prior to randomization.
14. Patients with previous or concomitant malignancy (not breast cancer) within the past 5 years EXCEPT adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix. Patients who have had a previous other malignancy must have been disease free for five years.
15. Patients with other non-malignant systemic diseases including uncontrolled infections, uncontrolled type 2 diabetes mellitus, uncontrolled thyroid dysfunction, cardiovascular, renal, hepatic, and lung diseases which would prevent prolonged follow-up. Patients with previous history of thrombosis or thromboembolism can be included only if medically suitable. Patients with a known history of HIV are excluded.
16. Uncontrolled seizure disorders associated with falls.
17. Patients with abnormal renal function as evidenced by a serum creatinine equal to or greater than 3 mg/dL (265.2 mmol/L).
18. History of diseases with influence on bone metabolism, such as Paget's disease, Osteogenesis Imperfecta, and primary or secondary hyperthyroidism within 12 months prior to study entry.
19. Patients with baseline lumber spine or total hip BMD T-score below -2.0 SD.
20. Patients treated with systemic investigational drug(s) and/or device(s) within the past 30 days or topical investigational drugs within the past 7 days.

Additional Exclusion Criteria: (for Spine DXA)

* History of surgery at the lumbosacral spine, with or without implantable devices.
* Scoliosis with a Cobb angle >15 degree at the lumbar spine.
* Immobility, hyperostosis or sclerotic changes at the lumbar spine, or evidence of sclerotic abdominal aorta sufficient to interfere with DXA scan.
* Any disease of the spine that would preclude the proper acquisition of a lumbar spine DXA.

Additional protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2002-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, MD, Study Director — Novartis Pharmaceuticals
Locations (44):
- United States (43):
  - Highlands Oncology Group, Springdale, Arkansas
  - East Valley Hematology & Oncology, Burbank, California
  - Louisiana Oncology Associates, Lafayette, California
  - Wilshire Oncology Medical Group, LaVerne, California
  - Pacific Shores Medical Group, Long Beach, California
  - Clinical Trials & Research Associates, Inc., Montebello, California
  - Redwood Regional Medical Group, Santa Rosa, California
  - Cancer and Blood Institute of the Desert, Rancho Mirage, Colorado
  - Eastern Connecticut Hematology/Oncology Associates, Norwich, Connecticut
  - FL Community Cancer Center, Brooksville, Florida
  - Robert R. Carroll, MD, PA, Gainesville, Florida
  - Oncology Hematology Group of South Florida, Miami, Florida
  - Pasco Pinellas Cancer Center, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Research Network, Inc., Plantation, Florida
  - Bay Area Oncology, Tampa, Florida
  - Space Coast Medical, Titusville, Florida
  - Elmhurst Memorial Hospital, Elhurst, Illinois
  - Kentuckiana Cancer Institute, Louisville, Kentucky
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - New England Hematology/Oncology Associates, Wellesley, Massachusetts
  - Cook Research Department at Spectrum Health, Grand Rapids, Michigan
  - Metro Minnesota CCOP, Saint Louis Park, Minnesota
  - Hematology-Oncology Centers of the Northern Rockies, PC, Billings, Montana
  - Methodist Cancer Center, Omaha, Nebraska
  - Hematology-Oncology Associates of Northern NJ, Morristown, New Jersey
  - New Mexico Oncology Hematology, Ltd., Albuquerque, New Mexico
  - Hemoncare PC, Brooklyn, New York
  - Odyssey Research Services, Bismarck, North Dakota
  - Nashat Y. Gabrail MD Inc., Canton, Ohio
  - Oncology Partners Network, Cincinnati, Ohio
  - Physician Associates, Inc., Cincinnati, Ohio
  - Dayton Clinical Oncology Program, Dayton, Ohio
  - University of Pittsburgh Cancer Institute/Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology, Charleston, South Carolina
  - The Sarah Cannon Cancer Center, Nashville, Tennessee
  - St. Joseph Regional Cancer Center, Bryan, Texas
  - Cancer Specialists of South Texas, Corpus Christi, Texas
  - Center for Oncology Research & Tx. PA, Dallas, Texas
  - Northern Virginia Oncology Group, Fairfax, Virginia
  - Virginia Physicians, Inc.- Oncology, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Rockwood Clinic, PS, Spokane, Washington
- VA Medical Center, San Juan, Puerto Rico

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 602 participants (301 in the upfront arm and 301 in the delayed-start arm) were randomized. Of these, 600 participants (300 in each arm) were treated. One participant in the upfront arm withdrew before taking any study drug and one participant in the delayed-start arm withdrew for administrative reasons prior to taking any study drug.
Groups:
- Zoledronic Acid Upfront: Participants in the upfront arm received Zoledronic Acid 4 mg i.v. on Day 1 and every 6 months until disease progression (recurrence) or the end of study. Participants also received Letrozole 2.5 daily plus calcium (1000-1200 mg) and vitamin D (400-800 IU) daily.
  Letrozole : Participants received 2.5 mg daily.
  Zoledronic Acid : Participants received Zoledronic Acid 4 mg IV 15-minute infusion every 6 months.
- Zoledronic Acid Delayed-start: In lieu of a placebo arm, which was considered unethical for this trial, a delayed start arm was used. Participants who met certain clinical criteria indicating risk of lumbar spine or total hip fracture, or experienced clinical fracture unrelated to trauma or any asymptomatic fracture discovered at the Month 36 scheduled visit, were started on zoledronic acid 4 mg i.v. and for every 6 months until disease progression (recurrence) or end of study. Participants also received Letrozole 2.5 daily plus calcium (1000-1200 mg) and vitamin D (400-800 IU) daily.
  Letrozole : Participants received 2.5 mg daily.
  Zoledronic Acid : Participants received Zoledronic acid 4 mg IV 15-minute infusion every 6 months.
Period: Overall Study
Arm/Group | Zoledronic Acid Upfront | Zoledronic Acid Delayed-start
Started | 301 | 301
Intent-to-treat Population | 300 | 300
Completed | 180 | 175
Not Completed | 121 | 126
Not completed — Adverse Event | 41 | 46
Not completed — Abnormal laboratory value(s) | 1 | 1
Not completed — Abnormal test procedure results | 0 | 1
Not completed — Lack of Efficacy | 16 | 21
Not completed — Participant condition no longer required | 1 | 0
Not completed — Protocol Violation | 4 | 10
Not completed — Withdrawal by Subject | 34 | 26
Not completed — Lost to Follow-up | 7 | 9
Not completed — Administrative problems | 10 | 6
Not completed — Death | 7 | 4
Not completed — Unknown - Reason is missing | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Zoledronic Acid Upfront: Participants in the upfront arm received Zoledronic Acid 4 mg i.v. on Day 1 and every 6 months until disease progression (recurrence)or the end of study. Participants also received Letrozole 2.5 daily plus calcium (1000-1200 mg) and vitamin D (400-800 IU) daily.
  Letrozole : Participants received 2.5 mg daily.
  Zoledronic Acid : Participants received Zoledronic Acid upfront 4 mg IV 15-minute infusion every 6 months.
- Zoledronic Acid Delayed-start: In lieu of a placebo arm, which was considered unethical for this trial, a delayed start arm was used. Participants who met certain clinical criteria indicating risk of lumbar spine or total hip fracture, or experienced clinical fracture unrelated to trauma or any asymptomatic fracture discovered at the Month 36 scheduled visit, were started on Zoledronic Acid 4 mg i.v. and for every 6 months until disease progression (recurrence) or end of study. Participants also received Letrozole 2.5 daily plus calcium (1000-1200 mg) and vitamin D (400-800 IU) daily.
  Letrozole : Participants received 2.5 mg daily.
  Zoledronic Acid : Participants received Zoledronic Acid upfront 4 mg IV 15-minute infusion every 6 months.
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid Upfront | Zoledronic Acid Delayed-start | Total
Number analyzed (Participants) | 301 | 301 | 602
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (9.28) | 61.0 (8.92) | 61.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 301 | 301 | 602
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine (L1-L4) Bone Mineral Density (BMD)
Description: Bone mineral density (BMD) measurements were assessed by dual energy x-ray absorptiometry (DXA). The DXA devices of participating sites were cross-calibrated and the DXA results were compiled and analyzed by a central reader. Percent change = 100*((BMD at Month 12 - Baseline BMD)/Baseline BMD)). Missing data at month 12 were imputed by using the last observation carried forward (LOCF) method. Post-baseline non-missing data from month 6 were carried forward to month 12. Data prior to month 6 were not carried forward.
Time Frame: Baseline, 12 months
Population: Intent to treat (ITT population) was used. The ITT population contained all patients in the safety population for whom at least one post-baseline efficacy measurement was collected.
Measure: Mean (Standard Deviation); unit: Percentage of BMD
Groups:
- Zoledronic Acid Upfront: Participants in the upfront arm received Zoledronic Acid 4 mg i.v. on Day 1 and every 6 months until disease progression (recurrence)or the end of study. Participants also received Letrozole 2.5 daily plus calcium (1000-1200 mg) and vitamin D (400-800 IU) daily.
  Letrozole : Participants received 2.5 mg daily.
  Zoledronic Acid : Participants received Zoledronic Acid 4 mg IV 15-minute infusion every 6 months.
Arm/Group | Zoledronic Acid Upfront | Zoledronic Acid Delayed-start
Number analyzed (Participants) | 253 | 256
Percentage of BMD | 1.955 (3.3658) | -2.325 (3.9542)

2. Secondary Outcome: Percent Change From Baseline in Lumbar Spine (L1-L4) BMD
Description: Bone mineral density (BMD) measurements were assessed by dual energy x-ray absorptiometry (DXA). The DXA devices of participating sites were cross-calibrated and the DXA results were compiled and analyzed by a central reader.
  Percent change = 100*((BMD at Time Frame - Baseline BMD)/Baseline BMD)). Missing data beyond month 12 were not imputed by LOCF.
Time Frame: Baseline, 2 years, 3 years, 5 years
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percentage of BMD
Groups:
- Zoledronic Acid Delayed Start: In lieu of a placebo arm, which was considered unethical for this trial, a delayed start arm was used. Participants who met certain clinical criteria indicating risk of lumbar spine or total hip fracture, or experienced clinical fracture unrelated to trauma or any asymptomatic fracture discovered at the Month 36 scheduled visit, were started on Zoledronic Acid 4 mg i.v. and for every 6 months until disease progression (recurrence) or end of study. Participants also received Letrozole 2.5 daily plus calcium (1000-1200 mg) and vitamin D (400-800 IU) daily.
  Letrozole : Participants received 2.5 mg daily.
  Zoledronic Acid : Participants received Zoledronic Acid 4 mg IV 15-minute infusion every 6 months.
Arm/Group | Zoledronic Acid Upfront | Zoledronic Acid Delayed Start
Number analyzed (Participants) | 300 | 300
Percentage of BMD
  2 years (n=206,202) | 3.137 (4.1599) | -2.889 (5.0783)
  3 years (n=189,190) | 3.853 (4.5414) | -2.990 (5.7925)
  5 years (n=140,132) | 6.192 (5.9723) | -2.418 (7.4545)

3. Secondary Outcome: Percent Change From Baseline in Total Hip BMD
Description: Bone mineral density (BMD) measurements were assessed by dual energy x-ray absorptiometry (DXA). The DXA devices of participating sites were cross-calibrated and the DXA results were compiled and analyzed by a central reader.
  Percent change = 100*((BMD at Time Frame - Baseline BMD)/Baseline BMD)). Missing data at month 12 were imputed by using the LOCF method. Post-baseline non-missing data from month 6 were carried forward to month 12. Data prior to month 6 were not carried forward.
Time Frame: Baseline, 12 months, 2 years, 3 years, 5 years
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percentage of BMD
Arm/Group | Zoledronic Acid Upfront | Zoledronic Acid Delayed Start
Number analyzed (Participants) | 300 | 300
Percentage of BMD
  12 months (n=253,256) | 1.256 (2.5878) | -1.883 (3.3007)
  2 years (n=208,200) | 1.413 (2.9178) | -3.150 (4.0450)
  3 years (n=187,189) | 1.676 (3.6979) | -3.463 (5.2585)
  5 years (n=141,132) | 2.571 (4.8794) | -4.115 (6.1071)

4. Secondary Outcome: Percent Change From Baseline in Biochemical Markers of Bone Turnover, Serum N-Telopeptide (sNTX) and Bone-specific Alkaline Phosphatase (BSAP)
Description: Blood samples from a subset of participants (231 participants in total) were collected to measure the sNTX and BSAP. Missing data at month 12 were imputed by using the LOCF method. Post-baseline non-missing data from months 6 and 9 were carried forward to month 12. Data prior to month 6 were not carried forward. Missing data beyond month 12 were not imputed by LOCF.
Time Frame: Baseline, 12 months, 2 years, 3 years, 5 years
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percentage of biochemical markers
Arm/Group | Zoledronic Acid Upfront | Zoledronic Acid Delayed Start
Number analyzed (Participants) | 300 | 300
Percentage of biochemical markers
  sNTX, 12 months (n=87,85) | -20.1 (42.1) | 21.7 (55.2)
  sNTX, 2 years | NA (NA) — After data analysis was performed for the 24 month interim analysis, a technical problem with the sNTX assay was identified. As a result, sNTX data collected at time points after 12 months were not considered reliable for inclusion. | NA (NA) — After data analysis was performed for the 24 month interim analysis, a technical problem with the sNTX assay was identified. As a result, sNTX data collected at time points after 12 months were not considered reliable for inclusion.
  sNTX, 3 years | NA (NA) — After data analysis was performed for the 24 month interim analysis, a technical problem with the sNTX assay was identified. As a result, sNTX data collected at time points after 12 months were not considered reliable for inclusion. | NA (NA) — After data analysis was performed for the 24 month interim analysis, a technical problem with the sNTX assay was identified. As a result, sNTX data collected at time points after 12 months were not considered reliable for inclusion.
  sNTX, 5 years | NA (NA) — After data analysis was performed for the 24 month interim analysis, a technical problem with the sNTX assay was identified. As a result, sNTX data collected at time points after 12 months were not considered reliable for inclusion. | NA (NA) — After data analysis was performed for the 24 month interim analysis, a technical problem with the sNTX assay was identified. As a result, sNTX data collected at time points after 12 months were not considered reliable for inclusion.
  BSAP, 12 months (n=88,90) | -7.8 (28.2) | 19.0 (39.2)
  BSAP, 2 years (n=63,60) | -12.0 (26.3) | 19.9 (48.1)
  BSAP, 3 years (n=59,52) | -12.4 (23.2) | 10.6 (42.2)
  BSAP, 5 years (n=95,102) | -6.4 (35.4) | 11.9 (41.0)

5. Secondary Outcome: Incidence Rate of All Clinical Fractures
Description: The number of participants who experienced a clinical fracture at month 36 was assessed. Initial x-ray (both AP and lateral views) of the lumbar and thoracic spine were performed at baseline to exclude participants with evidence of fracture. In addition, repeated bone scan and/or x-ray were performed at the Principal Investigator's discretion during the course of the study to confirm evidence of clinical fracture, or at month 36 if there was no evidence of clinical fracture (lumbar and thoracic spine - lateral view). X-ray films were sent to a central reader.
Time Frame: 3 years
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid Upfront | Zoledronic Acid Delayed Start
Number analyzed (Participants) | 300 | 300
Participants | 18 | 21

6. Secondary Outcome: Time to Disease Recurrence/Relapse
Description: The median time to disease progression was assessed by Kaplan-Meier analysis. The Principal Investigator assessed each participant for disease recurrence at each visit. Further testing was performed at the discretion of the Principal Investigator and as clinically indicated. Disease progression was defined as chest wall and/or regional recurrence confirmed by positive cytology or biopsy, and/or distance recurrence of the 1) skin, subcutaneous tissue, and lymph nodes (other than local or regional), 2) bone marrow, 3) lung, 4) skeleton 5) liver and 6) central nervous system confirmed by positive cytology, biopsy, aspirate or radiology as appropriate.
Time Frame: over 5 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zoledronic Acid Upfront | Zoledronic Acid Delayed Start
Number analyzed (Participants) | 300 | 300
months | NA [NA to NA] — The median time to disease recurrence relapse was not achieved because of the small number of patients with recurrence. | NA [NA to NA] — The median time to disease recurrence relapse was not achieved because of the small number of patients with recurrence.

7. Secondary Outcome: Rate of Change From Baseline in Lumbar Spine (L1-L4) BMD
Description: The rate of change from baseline in BMD was assessed.
Time Frame: Baseline, 5 years
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: g/sq cm/month
Arm/Group | Zoledronic Acid Upfront | Zoledronic Acid Delayed Start
Number analyzed (Participants) | 300 | 300
g/sq cm/month | 0.01043 [0.00810 to 0.01277] | -0.00157 [-0.00396 to 0.00081]

8. Secondary Outcome: Rate of Change From Baseline in Total Hip BMD
Description: The rate of change from baseline in BMD was assessed.
Time Frame: Baseline, 5 years
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: g/sq. cm/month
Arm/Group | Zoledronic Acid Upfront | Zoledronic Acid Delayed Start
Number analyzed (Participants) | 300 | 300
g/sq. cm/month | 0.00226 [0.00071 to 0.00382] | -0.00625 [-0.00784 to -0.00466]

ADVERSE EVENTS:
Description: Overall, 602 participants (301 in the upfront arm and 301 in the delayed-start arm) were randomized. Of these, 600 participants (300 in each arm) were treated. One participant in the upfront arm withdrew before taking any study drug and one participant in the delayed-start arm withdrew for administrative reasons prior to taking any study drug.
Groups:
- Zoledronic Acid Upfront: Participants in the upfront arm received Zoledronic Acid 4 mg i.v. on Day 1 and every 6 months until disease progression (recurrence)or the end of study. Participants also received Femara 2.5 daily plus calcium (1000-1200 mg) and vitamin D (400-800 IU) daily.
  Letrozole : Participants received 2.5 mg daily. Zoledronic Acid : Participants received Zoledronic Acid 4 mg IV 15-minute infusion every 6 months.
Arm/Group | Zoledronic Acid Upfront | Zoledronic Acid Delayed-start
Serious Adverse Events (participants affected / at risk) | 83/300 | 71/300
Other Adverse Events (participants affected / at risk) | 283/300 | 275/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid Upfront (N=300) | Zoledronic Acid Delayed-start (N=300)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 2 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 4
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiomyopathy acute (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 4
Coronary artery occlusion (Cardiac disorders) | 0 | 4
Coronary artery stenosis (Cardiac disorders) | 1 | 2
Dilatation ventricular (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 2 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Oesophageal mass (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 4 | 2
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 3
Arthritis bacterial (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 1 | 0
Breast cellulitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 1 | 1
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 3
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Skin bacterial infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Urosepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Breast injury (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Device breakage (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 10 | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Bone density decreased (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 9
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Degeneration of uterine fibroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 3
Dementia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0
Subdural hygroma (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 2
Ovarian cyst (Reproductive system and breast disorders) | 1 | 2
Rectocele (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 4
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Jugular vein distension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid Upfront (N=300) | Zoledronic Acid Delayed-start (N=300)
Anaemia (Blood and lymphatic system disorders) | 13 | 20
Constipation (Gastrointestinal disorders) | 29 | 28
Diarrhoea (Gastrointestinal disorders) | 25 | 31
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 | 15
Nausea (Gastrointestinal disorders) | 39 | 40
Chest pain (General disorders) | 18 | 9
Fatigue (General disorders) | 101 | 88
Oedema peripheral (General disorders) | 36 | 30
Pain (General disorders) | 16 | 14
Pyrexia (General disorders) | 28 | 14
Bronchitis (Infections and infestations) | 17 | 6
Sinusitis (Infections and infestations) | 19 | 15
Upper respiratory tract infection (Infections and infestations) | 26 | 26
Urinary tract infection (Infections and infestations) | 37 | 26
Hypercholesterolaemia (Metabolism and nutrition disorders) | 21 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 141 | 136
Arthritis (Musculoskeletal and connective tissue disorders) | 22 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 44 | 52
Bone pain (Musculoskeletal and connective tissue disorders) | 48 | 24
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 17
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 17 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 33 | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 61 | 47
Neck pain (Musculoskeletal and connective tissue disorders) | 16 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45 | 40
Dizziness (Nervous system disorders) | 29 | 22
Headache (Nervous system disorders) | 39 | 37
Hypoaesthesia (Nervous system disorders) | 17 | 17
Paraesthesia (Nervous system disorders) | 17 | 6
Anxiety (Psychiatric disorders) | 24 | 25
Depression (Psychiatric disorders) | 35 | 42
Insomnia (Psychiatric disorders) | 41 | 29
Breast pain (Reproductive system and breast disorders) | 19 | 18
Vulvovaginal dryness (Reproductive system and breast disorders) | 24 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 38
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 25
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 18
Rash (Skin and subcutaneous tissue disorders) | 19 | 17
Hot flush (Vascular disorders) | 122 | 118
Hypertension (Vascular disorders) | 30 | 24
Lymphoedema (Vascular disorders) | 19 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.